CLINICAL TRIAL: NCT06152913
Title: All Hands on Deck: Youth, Therapists, Parents and School Professionals Joining Forces in a Personalized, Brief and Intensive Exposure-based Intervention for Youth With Persistent Anxiety or Obsessive Compulsive Disorder
Brief Title: HANDS-ON: a Personalized, Brief and Intensive Exposure-based Intervention for Youth With Persistent Anxiety or OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Accare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PSY-2223-S-0358
Record Dates: First submitted 2023-11-15; First posted 2023-12-01 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Anxiety Disorders; Obsessive-Compulsive Disorder; Obsessive-Compulsive Disorder in Children; Obsessive-Compulsive Disorder in Adolescence
Keywords: Anxiety; OCD; Non-responder; Exposure; Children and adolescents; CBT
MeSH Terms: conditions — Anxiety Disorders; Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Multiple baseline single-case experimental design
Masking Description: Note that research assistants will be blinded for the baseline length of participants during the interview assessments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HANDS-ON treatment with random baselines (Experimental): Participants are randomly allocated to one of four baseline periods (2.5 weeks, 3 weeks, 3.5 weeks, or 4 weeks). Participants then receive the HANDS-ON treatment. This treatment consists of three phases across nine weeks. After the treatment, there is a follow-up period of 4 weeks.
  Interventions: Behavioral: HANDS-ON treatment

INTERVENTIONS:
Behavioral: HANDS-ON treatment — The HANDS-ON treatment consists of three phases:
  Phase I (preparatory phase, 3 weeks) entails motivation for and commitment to treatment (including meaning in life), collaboration with parents and school professionals, setting individual treatment goals, preparing related exposure exercises. Phase II (intensive phase, 4 weeks) contains intensive, therapist-assisted exposure in a child's natural environment. Phase III (consolidation, 2 weeks) consists of continuation of exposure and consolidation. In this phase, there are weekly sessions with the therapist.

SUMMARY:
A substantial part of children/adolescents with anxiety or obsessive-compulsive disorder (AD/OCD) do not profit substantially from first-choice treatment (i.e., cognitive behavioral therapy; CBT). For them, no evidence-based treatment is available. The aim of this project is to evaluate and optimize a newly-developed personalized, short, and intensive exposure-based intervention, 'HANDS-ON', for 'treatment non-responders'. Collaboration with children, parents and teachers, guided exposure in a child's natural environment, personalized treatment goals and meaning/motivation are central principles.

Methods: A multiple baseline single-case experimental design is used (qualitative and quantitative). Participants are children/adolescents (10-18 years; N=12) with an AD/OCD diagnosis for whom standard CBT did not lead to sufficient improvement. Children and parents are asked to complete questionnaires before, during, and after the treatment. Children, parents, and school professionals will be asked to participate in qualitative interviews to evaluate their experiences with the HANDS-ON treatment program.

DETAILED DESCRIPTION:
BACKGROUND Nearly half of children and adolescents with anxiety or obsessive-compulsive disorders do not reach remission after first-choice treatment (cognitive behavioral therapy; CBT) and 10-25% discontinue treatment prematurely. For them, no evidence-based treatment is available. They may have severe symptoms with a huge impact on daily functioning, quality of life, family life, and society. These youth are at risk of developmental delays, among others due to school refusal. They often receive time-consuming, expensive treatment without evidence of effectiveness.

OBJECTIVES The aim of this project is to evaluate and optimize a newly-developed treatment for this group. This treatment, 'HANDS-ON', is innovative, short and intensive, based on scientific research and insights from clinical practice. Collaboration with children, parents and teachers, guided exposure in a child's natural environment, personalized treatment goals and meaning/motivation are central principles.

Our research questions are:

1. Quantitative: What are (within-subjects) effects of HANDS-ON on personalized goal attainment, anxiety/OCD severity, and functioning in youth with persistent AD/OCD?
2. Qualitative: What are the experiences, facilitators and barriers of HANDS-ON from a child, parent, school professional and therapist perspective?

The results of this study will be used to improve HANDS-ON, with the aim to further investigate its effectiveness in a randomised controlled trial as a next step.

METHOD Participants are 12 children/adolescents with persistent anxiety- or obsessive-compulsive symptoms (treatment non-responders). Inclusion criteria: a) age 10-18 years; b) diagnosis of anxiety disorder or obsessive-compulsive disorder (DSM-5); c) non-response to previous CBT (CBT with insufficient effect). Co-morbid diagnoses are allowed except for those interfering with safety or warranting immediate treatment (e.g., acute suicidality or psychosis).

Design: multiple baseline single-case experimental design. Participants will be randomised to one of four baseline periods (2.5-4 weeks), followed by HANDS-ON (9 weeks) and follow-up (4 weeks). Progress on personalized treatment goals (primary outcome) and on symptoms (impairment and avoidance, secondary outcome) will be measured daily. Other outcomes will be measured at baseline (T0), start HANDS-ON (T1, subset), after HANDS-ON (T2), and at follow-up (T3). Semi-structured interviews (qualitative evaluation) will be conducted with the youth, their parents, school professionals, and therapists (post-treatment).

Analyses: The primary outcome will be analysed using randomisation tests and combined using meta-analytic analyses. Descriptive analyses and tests for repeated measures will be used to analyse secondary outcomes. Qualitative interviews will be recorded and analysed using thematic text analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 10-18 years old;
* Meeting DSM-5 criteria for an anxiety disorder/OCD, based on a semi-structured interview (SCID-5 Jr; [12]) and clinical judgement of an experienced and authorized clinician;
* Non-responder to previous CBT (insufficient benefits from previous CBT for AD/OCD).

Comorbid diagnoses are allowed except for those interfering with safety or warranting immediate treatment, e.g., acute suicidality or psychosis.

Exclusion Criteria:

* Severe psychiatric symptoms other than anxiety/OCD interfering with safety or warranting immediate intervention, e.g. psychosis or acute suicidality.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Individualized treatment goals | Daily child ratings (13 weeks), Timepoint0 (start baseline), Timepoint1 (pre-treatment), Timepoint2 (post-treatment, 9 weeks later), and Timepoint3 (follow-up, 4 weeks later); parent-rating at Timepoint0, Timepoint1, Timepoint2 and Timepoint3
  Measured daily using the Goal Based Outcomes (GBO) questionnaire. Each participant will set 3 individualized anxiety/OCD-related goals for the treatment, scored on a scale from 1 - 10, where higher scores indicate improved goal progress.

SECONDARY OUTCOMES:
Severity/remission of primary diagnosis | Child and parent ratings at Timepoint0 (start baseline), Timepoint2 (post-treatment, 9 weeks after Timepoint1 [pre-treatment, 2.5-4 weeks after start baseline]), and Timepoint3 (follow-up, 4 weeks after Timepoint2)
  Measured using the Structured Clinical Interview for DSM-5 Childhood Disorders (SCID-5 Junior) [child and parent report], with severity indicated as Clinical Severity Rating rated from 1 - 8 (adapted from the Anxiety Disorders Interview Schedule for DSM-IV, ADIS-IV) and higher ratings indicating higher severity.
Anxiety symptoms | Child and parent ratings at Timepoint0 (start baseline), Timepoint1 (pre-treatment, 2.5-4 weeks after start baseline), Timepoint2 (post-treatment, 9 weeks after Timepoint1), Timepoint3 (follow-up, 4 weeks after Timepoint2)
  Measured using the Revised Child Anxiety and Depression Scale (RCADS) [child and parent report], with items rated as 0 ('Never'), 1 ('Sometimes'), 2 ('Often'), and 3 ('Always') and higher scores indicating more severity.
OCD severity | Combined child and parent ratings at Timepoint0 (start baseline), Timepoint1 (pre-treatment, 2.5-4 weeks after start baseline), Timepoint2 (post-treatment, 9 weeks after Timepoint1), Timepoint3 (follow-up, 4 weeks after Timepoint2)
  Only in case of OCD. Measured using the Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) [combined child and parent report], with items rated from 0 - 4 and higher scores indicating more severity.
Family accommodation | Parent ratings at Timepoint0 (start baseline), Timepoint2 (post-treatment, 9 weeks after Timepoint1 [pre-treatment, 2.5-4 weeks after start baseline]), and Timepoint3 (follow-up, 4 weeks after Timepoint2)
  Measured using the Family Accommodation Scale - Anxiety/OCD (FASA, parent version), with items rated from 0 - 4 and higher scores indicating more family accommodation.
School refusal | Child and parent ratings at Timepoint0 (start baseline), Timepoint2 (post-treatment, 9 weeks after Timepoint1 [pre-treatment, 2.5-4 weeks after start baseline]), and Timepoint3 (follow-up, 4 weeks after Timepoint2)
  Measured using the School Refusal Assessment Scale-Revised for Children (SRAS-R(-NL)-C/P) [child and parent report], with items ranging from 0 - 6 and higher scores indicating more school refusal.
Motivation | Child ratings at Timepoint0 (start baseline), Timepoint1 (pre-treatment, 2.5-4 weeks after start baseline), Timepoint2 (post-treatment, 9 weeks after Timepoint1), Timepoint3 (follow-up, 4 weeks after Timepoint2)
  Measured using three items with self-developed visual analogue slider scales, with ratings ranging from 0 - 100 and higher scores indicating more motivation.
Clinical global impression | Clinician ratings at Timepoint0 (start baseline), Timepoint1 (pre-treatment, 2.5-4 weeks after start baseline), Timepoint2 (post-treatment, 9 weeks after Timepoint1), Timepoint3 (follow-up, 4 weeks after Timepoint2)
  Measured using the Clinical Global Impression (CGI) Scale (Severity, Improvement) [clinician rated], with two items ranging from 1 - 7 and higher scores indicating more deterioration.
Treatment adherence | Clinician rating at Timepoint2 (post-treatment, 9 weeks after Timepoint1 [pre-treatment] and 11.5-13 weeks after Timepoint0 [pre-baseline])
  Checklist for therapists [clinician rated], with checkboxes indicating adherence (or deviations) to treatment components
Qualitative interview | Between Timepoint2 (post-treatment, 9 weeks after Timepoint1 [pre-treatment] and 11.5-13 weeks after Timepoint0 [pre-baseline]) and Timepoint3 (follow-up, 4 weeks after Timepoint2)
  Treatment evaluation, child, parent, and therapist interviews
Treatment satisfaction questionnaire | Child and parent ratings at Timepoint2 (post-treatment, 9 weeks after Timepoint1 [pre-treatment] and 11.5-13 weeks after Timepoint0 [pre-baseline])
  Measured using a self-developed satisfaction scale [child and parent reports], scale title and minimum/maximum values to be specified
Daily anxiety or OCD symptoms | Child rating daily through baseline (2.5-4 weeks), treatment (9 weeks) and partially during follow-up (91 days [13 weeks] for each participant)
  Measured daily using two self-developed visual analogue slider scales. One slider measures impairment on a scale from 0 - 100. The other measures avoidance on a scale from 0 - 100. Higher scores indicate more impairment and avoidance.

OTHER OUTCOMES:
Descriptive measures at baseline | Timepoint0 (start baseline)
  Age in years
Descriptive measures at baseline | Timepoint0 (start baseline)
  Gender
Descriptive measures at baseline | Timepoint0 (start baseline)
  DSM-5 classification (primary diagnosis, co-morbid diagnoses)
Descriptive measures at baseline | Timepoint0 (start baseline)
  Educational level
Descriptive measures at baseline | Timepoint0 (start baseline)
  Family composition
Descriptive measures at baseline | Timepoint0 (start baseline)
  Year of onset anxiety or OCD
Descriptive measures at baseline | Timepoint0 (start baseline)
  Previous treatment

CONTACTS AND LOCATIONS:
Overall Officials: L. Wolters, Dr., Principal Investigator — Accare; M. H. Nauta, Dr., Study Chair — Accare, University of Groningen
Locations (1):
- Accare, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
After completion of the present study, data can be made available and shared for re-use and participants will be asked informed consent for this (Findable, Accessible, Interoperable, and Reusable ['FAIR'] data). Requests for data sharing will be assessed by the Principal investigator. When data sharing is requested, an agreement will be drawn up. Consent is asked for using and sharing pseudonymized data for instance for reviews, (individual patient data) meta-analyses, and questionnaire (validation) studies.
  The pseudonymized merged, prepared and analysed dataset may become available for re-use, in line with the FAIR principles. Since the data is sensitive, data will not be openly and publicly available. However, they could be shared for research purposes such as for (individual patient data) meta-analyses, and questionnaire (validation) studies by established experts in the field. The Principle Investigator is responsible for the data and can be contacted for questions.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data can be requested after publication.
Access Criteria: The pseudonymized merged, prepared and analysed dataset may become available for re-use, in line with the FAIR principles. Since the data is sensitive, data will not be openly and publicly available. However, they could be shared for research purposes such as for (individual patient data) meta-analyses, and questionnaire (validation) studies by established experts in the field. The Principle Investigator is responsible for the data and can be contacted for questions.

REFERENCES:
- [Background] Law, D., & Jacob, J. (2015). Goals and Goal Based Outcomes (GBOs): Some useful information. Third Edition. London, UK: CAMHS Press
- [Background] Wante, Braet, C., Bögels, S., & Roelofs, J. (2021). SCID-5 Junior: Een semi-gestructureerd klinisch interview voor DSM-5 stoornissen bij kinderen en adolescenten. Boom. http://hdl.handle.net/1854/LU-8695564
- [Background] Chorpita BF, Yim L, Moffitt C, Umemoto LA, Francis SE. Assessment of symptoms of DSM-IV anxiety and depression in children: a revised child anxiety and depression scale. Behav Res Ther. 2000 Aug;38(8):835-55. doi: 10.1016/s0005-7967(99)00130-8. PMID 10937431
- [Background] Scahill L, Riddle MA, McSwiggin-Hardin M, Ort SI, King RA, Goodman WK, Cicchetti D, Leckman JF. Children's Yale-Brown Obsessive Compulsive Scale: reliability and validity. J Am Acad Child Adolesc Psychiatry. 1997 Jun;36(6):844-52. doi: 10.1097/00004583-199706000-00023. PMID 9183141
- [Background] Lebowitz ER, Woolston J, Bar-Haim Y, Calvocoressi L, Dauser C, Warnick E, Scahill L, Chakir AR, Shechner T, Hermes H, Vitulano LA, King RA, Leckman JF. Family accommodation in pediatric anxiety disorders. Depress Anxiety. 2013 Jan;30(1):47-54. doi: 10.1002/da.21998. Epub 2012 Sep 10. PMID 22965863
- [Background] Heyne, D. A., Vreeke, L., & Maric, M. (2008). School Refusal Assessment Scale-Revised (kindversie) Nederlandse vertaling en bewerking. Universiteit Leiden. https://effectivechildtherapy.fiu.edu/pluginfile.php/1783/mod_resource/content/2/41_School%20Refusal%20Scale.pdf.pdf